CLINICAL TRIAL: NCT00336518
Title: Efficacy and Safety of Continuing for a Total of 48 or Prolonging for a Total of 72 Weeks of Combined Treatment of Patients Receiving Pegasys and Copegus Who Are Biochemical Responders But Virological Non-Responders at Week 12 or Week 24
Brief Title: Continuing Treatment With Pegasys and Copegus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Májbetegekért Alapítvány (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBA 1/2005; ML 20142; EuDract: 2005-004531-22
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2006-06-13 (Estimated); Status verified 2005-08

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

INTERVENTIONS:
Drug: peginterferon alfa-2a
Drug: ribavirin

SUMMARY:
Primary objective is to measure sustained viral response given to continuation or prolongation of combined Pegasys&Copegus treatment

Secondary objective is to measure histological response given to continuation or prolongation of combined Pegasys&Copegus treatment measured by non-invasive methods

DETAILED DESCRIPTION:
Prospective, multicentre, randomized, open-label comparative study

According to our national guideline of management of patient with chronic viral hepatitis, patients need to stop therapy if they do not achieve response.

These patients can enter to the study at two time points:

* at week 16, if HCV RNS PCR measured at week 12 is positive and serum ALT > 1ULN, but decreased
* at week 28, if HCV RNS PCR measured at week 24 is still positive, but serum ALT < 2ULN.

Patients are randomized to one of the following arms:

* S (standard) group: Pegasys&Copegus combined therapy 180 mcg/week & weight/based 1000-1200 mg/day for a total of 48 weeks of treatment
* P (prolonged) group: Pegasys&Copegus combined therapy 180 mcg/week & -weight/based 1000-1200 mg/day for a total of 72 weeks of treatment.

After completing treatment period patients enter into a 24-week follow up.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients above 18 and below 65 years of age chronically infected with genotype 1 HCV receiving combined Pegasys&Copegus treatment first time in-line with the valid treatment guideline approved by the National Interferon Committee (see attached guideline)

Subgroup 1:

* Positive HCV PCR result at week 12 of the ongoing treatment
* ALT > 1ULN, but the value decreased by week 12

Subgroup 2:

* ALT was normal and PCR was positive at week 12, therefore combined treatment could be continued between week 12 and 24 based on the approved guideline
* Positive HCV RNA PCR at week 24 of the ongoing treatment
* GPT < 2 ULN at week 24 of the ongoing treatment.

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Therapy with any systemic anti-neoplastic or immunomodulatory treatment at inclusion or within 6 months prior to it
* Any investigational drug usage at inclusion or within 6 weeks prior to it
* Co/infection with hepatitis A, B or HIV
* Any chronic liver disease other than HCV infection
* Sign or symptom of hepatocellular carcinoma
* Decompensated liver disease
* History of depression or any other relevant psychiatric disease which, in the opinion of a psychiatrist or neurologist, contraindicates study therapy
* Uncontrolled thyroid dysfunction
* Severe retinopathy
* Evidence of regular alcohol consumption at inclusion or within 1 year prior to it
* Any side effect probably caused by ongoing combined treatment which, in the opinion of the investigator, contraindicates continuation of the therapy or necessitates dose reduction of any drug in the combination therapy
* Unwillingness to provide informed consent

Subgroup 1:

Laboratory findings at week 16 of the ongoing combined Pegasys&Copegus treatment:

* ANC <1000/mm3
* PLT <75.000/mm3
* hemoglobin <10g/dl
* creatinine >1,5 ULN

Subgroup 2:

Laboratory findings at week 28 of the ongoing combined Pegasys&Copegus treatment:

* ANC <1000/mm3
* PLT <75.000/mm3
* hemoglobin <10g/dl
* creatinine >1,5 ULN

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-06; Study Completion 2009-07

PRIMARY OUTCOMES:
Sustained viral response given to continuation or prolongation of combined Pegasys&Copegus treatment

SECONDARY OUTCOMES:
Histological response given to continuation or prolongation of combined Pegasys&Copegus treatment measured by non-invasive methods

CONTACTS AND LOCATIONS:
Overall Officials: János Schuller, Dr., Principal Investigator — Májbetegekért Alapítvány
Locations (1):
- Szt. László Hospital, Budapest, Hungary